CLINICAL TRIAL: NCT02521948
Title: Clinical Study to Evaluate the Safety and Performance of MANTA Vascular Closure Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essential Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSD-051
Record Dates: First submitted 2015-08-07; First posted 2015-08-13 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-02

CONDITIONS: Femoral Arteriotomy Closure
Keywords: MANTA; Arterial Closure Device; Large Bore Closure Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MANTA Vascular Closure Device (Experimental): The MANTA device, developed by Essential Medical, Inc., is a vascular closure device (VCD) intended for use in catheterization laboratories following percutaneous cardiac or peripheral procedures that use the retrograde common femoral artery access route for large bore (10-18F) interventional devices.
  Interventions: Device: MANTA Vascular Closure Device

INTERVENTIONS:
Device: MANTA Vascular Closure Device — The MANTA device developed by Essential Medical, Inc., is a vascular closure device (VCD) intended for use in catheterization laboratories following percutaneous cardiac or peripheral procedures that use the retrograde common femoral artery access route for large bore (10-18F) interventional devices.

SUMMARY:
The purpose of this study is to evaluate the safety and performance of the MANTA Vascular Closure Device (VCD) to close the arteriotomy following percutaneous cardiovascular procedures utilizing large bore sheaths for purposes of supporting a CE Mark (Conformite Europeenne--"European Conformity") and other regulatory submissions. The study will assess whether the MANTA VCD is safe and performs as intended for large-bore vascular closure after interventional procedures.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and performance of MANTA in achieving hemostasis in femoral arterial access sites in patients undergoing percutaneous transcatheter interventional procedures using a 10-18F procedure sheath (such as Transcather Aortic Valve Replacement (TAVR), Balloon Aortic Valvuloplasty (BAV) and Endovascular Aneurysm Repair (EVAR)) for purposes of obtaining a CE Mark in the European Union.

The study will evaluate hemostasis success, time to hemostasis and ambulation, treatment success, and the rate of access-site-related complications in comparison to published literature on other hemostasis techniques for closing these large bore punctures (primarily, surgical closure and suture-mediated percutaneous closure.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for non-emergent transcatheter interventional procedure via a 10-18F femoral sheath (e.g., transcatheter aortic valve replacement [TAVR], balloon aortic valvuloplasty [BAV], Abdominal Aortic Aneurysm [AAA] stent-graft placement)
* Eligible for sheath removal in the catheterization lab
* Age ≥18 years
* Understand and sign the study specific written informed consent form
* Able and willing to fulfill the follow-up requirements
* In the Investigator's opinion, the patient is suitable for the MANTA vascular closure device, conventional hemostasis techniques and participation in an investigational trial
* Patients of childbearing age with Negative Pregnancy Test within 7 days of procedure

Exclusion Criteria:

Baseline Exclusions:

* Patients who are known to be pregnant or lactating
* Patients who are immunocompromised or with pre-existing autoimmune disease
* Patients who have a systemic infection or a local infection at or near the access site
* Patients requiring a re-puncture at a site previously punctured within 48 hours
* Patients with significant anemia (hemoglobin < 6.5 mmol/l, Hct<30)
* Patients who are morbidly obese or cachectic (BMI >40 or <20)
* Patients with Systolic Blood Pressure >180 mmHg, unless Systolic Pressure can be lowered by pharmacological agents prior to closure
* Patients who are currently participating in another clinical trial of an investigational device or drug that has not concluded the follow-up period
* Patients in whom an antegrade puncture is performed or planned
* Patients with a known bleeding disorder including thrombocytopenia (platelet count <150 x 10^9/L), thrombasthenia, hemophilia, or von Willebrand's disease
* Patients with a femoral artery <6 mm in diameter, femoral artery stenosis resulting in a vessel diameter <6 mm, or patients with severe peripheral vascular disease
* Common femoral artery with fluoroscopically visible calcium, as determined by Angio CT, precluding safe access in the opinion of the investigator
* Patients with allergy to bovine materials, collagen and/or collagen products, or polyglycolic or polylactic acid polymers
* Patients who cannot adhere to or complete the investigational protocol for any reason including but not limited to geographical residence or life threatening disease
* Patients with Sheehan Disability Scale (SDS) scores >12
* Patients punctured through a vascular graft
* Patients with known allergy to stainless steel or nickel
* Patients who have acute ST-elevation myocardial infarction within 48 hours prior to procedure
* Patients with unilateral or bilateral lower extremity amputation
* Patients with renal insufficiency (serum creatinine >2.5 mg/dl)
* Patients undergoing therapeutic thrombolysis
* Patients who are unable to ambulate at baseline
* Patients undergoing an interventional procedure whom are being treated with warfarin
* Patients requiring a continuous oral anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- San Raffaele Hospital, Milan, Italy
- Netherlands (2):
  - St. Antonius Ziekenhuis, Nieuwegein
  - Erasmus Medical Center, Rotterdam

REFERENCES:
- [Background] Ben-Dor I, Looser P, Bernardo N, Maluenda G, Torguson R, Xue Z, Lindsay J, Pichard AD, Satler LF, Waksman R. Comparison of closure strategies after balloon aortic valvuloplasty: suture mediated versus collagen based versus manual. Catheter Cardiovasc Interv. 2011 Jul 1;78(1):119-24. doi: 10.1002/ccd.22940. PMID 21681898
- [Background] Nelson PR, Kracjer Z, Kansal N, Rao V, Bianchi C, Hashemi H, Jones P, Bacharach JM. A multicenter, randomized, controlled trial of totally percutaneous access versus open femoral exposure for endovascular aortic aneurysm repair (the PEVAR trial). J Vasc Surg. 2014 May;59(5):1181-93. doi: 10.1016/j.jvs.2013.10.101. Epub 2014 Jan 17. PMID 24440678
- [Background] Kadakia MB, Herrmann HC, Desai ND, Fox Z, Ogbara J, Anwaruddin S, Jagasia D, Bavaria JE, Szeto WY, Vallabhajosyula P, Li R, Menon R, Kobrin DM, Giri J. Factors associated with vascular complications in patients undergoing balloon-expandable transfemoral transcatheter aortic valve replacement via open versus percutaneous approaches. Circ Cardiovasc Interv. 2014 Aug;7(4):570-6. doi: 10.1161/CIRCINTERVENTIONS.113.001030. Epub 2014 Jul 15. PMID 25027520

RESULTS

PARTICIPANT FLOW:
Groups:
- MANTA Vascular Closure Device (Total): The MANTA device, developed by Essential Medical, Inc., is a vascular closure device (VCD) intended for use in catheterization laboratories following percutaneous cardiac or peripheral procedures that use the retrograde common femoral artery access route for large bore (10-18F) interventional devices.
Period: Overall Study
Arm/Group | MANTA Vascular Closure Device (Total)
Started | 50
Completed | 37
Not Completed | 13
Not completed — Adverse Event | 2
Not completed — Death | 4
Not completed — Lost to Follow-up | 1
Not completed — Did not attend one or both follow-ups | 6

BASELINE CHARACTERISTICS:
Population: Total MANTA device population
Arm/Group | MANTA Vascular Closure Device (Total)
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 79.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Complications
Description: Composite endpoint that includes any of the following adverse events:
  * Access site-related bleeding requiring blood transfusion or vascular repair
  * Vascular injury requiring repair (e.g. perforation, dissection, arterio-venous fistula, retroperitoneal bleed, pseudoaneurysm)
  * Femoral artery stenosis at the access site requiring intervention
  * New ipsilateral lower extremity ischemia causing a threat to the viability of the limb
  * Access site-related infection requiring intravenous antibiotics and/or extended hospitalization
  * New onset access site-related neuropathy in the ipsilateral lower extremity requiring surgical repair
  * Permanent access site-related nerve injury (lasting>30 days)
Time Frame: Within either the first 30 days (plus or minus 7 days) after the procedure or the first 60 days (plus or minus 14 days) after the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | MANTA Vascular Closure Device (Total)
Number analyzed (Participants) | 50
Participants | 3

2. Primary Outcome: Hemostasis Success
Description: Hemostasis at the puncture site within 10 minutes of cutting the MANTA suture without need for manual or mechanical compression and without later re-bleeding (trivial or subcutaneous oozing will not be considered bleeding; light finger pressure to control subcutaneous oozing will not be considered manual compression)
Time Frame: Within the first 10 minutes of cutting the MANTA suture
Measure: Count of Participants; unit: Participants
Groups:
- 14F MANTA Device: 14F subgroup of MANTA device
- 18F MANTA Device: 18F subgroup of MANTA device
Arm/Group | MANTA Vascular Closure Device (Total) | 14F MANTA Device | 18F MANTA Device
Number analyzed (Participants) | 50 | 16 | 34
Participants | 47 | 16 | 31

3. Secondary Outcome: Time to Hemostasis
Description: The elapsed time between MANTA deployment (withdrawal of sheath from artery) and first observed and confirmed arterial hemostasis (no or minimal subcutaneous oozing and the absence of expanding or developing hematoma).
Time Frame: Time between MANTA deployment and first observed and confirmed arterial hemostasis up to ten (10) minutes after MANTA device is deployed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | MANTA Vascular Closure Device (Total)
Number analyzed (Participants) | 50
minutes | 2.38 (6.63)

ADVERSE EVENTS:
Time Frame: 60 days
Groups:
- Device Related Adverse Events: Device related adverse events for the overall population
Arm/Group | MANTA Vascular Closure Device (Total) | Device Related Adverse Events
All-Cause Mortality (participants affected / at risk) | 4/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 20/50 | 3/50
Other Adverse Events (participants affected / at risk) | 45/50 | 32/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MANTA Vascular Closure Device (Total) (N=50) | Device Related Adverse Events (N=50)
Excessive access site bleeding (Vascular disorders) | 2 | 2
Pseudoaneurysm (Vascular disorders) | 1 | 1
Bleeding/hemorrhage (Vascular disorders) | 2 | 0 — Not related to access site or MANTA
Infection (Infections and infestations) | 3 | 0 — Not related to access site/MANTA device
Other (Cardiac disorders) | 15 | 0
Minor Stroke (Nervous system disorders) | 1 | 0
Cerebrovascular Attack (Vascular disorders) | 1 | 0
Other (Gastrointestinal disorders) | 2 | 0
Other (Renal and urinary disorders) | 1 | 0
Other (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Other (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MANTA Vascular Closure Device (Total) (N=50) | Device Related Adverse Events (N=50)
Excessive access site bleeding (Vascular disorders) | 3 | 3
Hematoma >6cm (Vascular disorders) | 10 | 10
Hematoma <= 6cm (Vascular disorders) | 19 | 19
Pseudoaneurysm (Vascular disorders) | 0 | 0
Femoral artery stenosis at access site (Vascular disorders) | 17 | 17
Other (Cardiac disorders) | 30 | 0 — All other AEs

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No